CLINICAL TRIAL: NCT01432509
Title: DiabeNord: A 5-year Prospective Follow-up Cohort Study in Pre-diabetic Subjects for the Identification of New Biomarkers
Brief Title: Prospective Follow-up of a Cohort of Pre-diabetics in the North of France (DiabeNord)
Acronym: DiabeNord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC12_0385; ID-RCB Number : 2011-A00565-36 (Other: Afssaps - French Health Products Safety Agency)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Prediabetes
Keywords: Pre-diabetes; Type 2 diabetes; Biomarkers; Cohort; Diabetes Risk Score; Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperglycemia
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prediabetes screening and prospective follow-up over 5 years — The study period per patient is 5 years. The planned schedule of the study is as follows :
  * Enrollment at visit V0 of subjects at high metabolic risk, based on a biological value (within the past 2 months) of moderate fasting hyperglycaemia (blood glucose ≥ 1,10 g/l and < 1,26 g/l) or fasting blood glucose ≥ 1 g/l and < 1,10 g/l with HbA1c ≥ 6,5%.
  * First biological sample (B0) within 1 month following V0 (measuring fasting blood glucose + glycated hemoglobin HbA1c + lipid profile + creatinemia + liver function; and establishment of a biological sample collection to identify biomarkers).
  * Annual follow-up for five years consisting in one blood sample (B1 to B5) measuring the same parameters as V0 + biological sample collection, and questionnaire on major health events or health events related to study procedures.
  * End of study phone call

SUMMARY:
The purpose of this study is to identify in prediabetic subjects, physiopathological changes involved in the evolution to type 2 diabetes mellitus and to identify new biomarkers of type 2 diabetes risk in this population.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a real public health issue, with an exponential incidence. Before its diagnosis, several physiopathological changes are already taking place, such as insulin resistance of target tissues and the progressive inability of pancreatic beta cells to produce insulin. The objective of this study is a better understanding of the prediabetic stage and mechanisms involved in the possible development of T2D, by way of a five-year follow-up cohort study in 207 prediabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Previous history (within 2 months prior to enrollment visit) of fasting blood glucose ≥ 1,10 g/l and < 1,26 g/l OR fasting blood glucose ≥ 1 g/l and < 1,10 g/l with HbA1c ≥ 6,5%.

Exclusion Criteria:

* Fasting glycemia ≥ 1.26 g/l
* History of treatment with oral antidiabetics
* History of treatment with insulin, except gestational diabetes
* Subject with any history or presence of significant hematologic (coagulation, thrombopenia, …), hepatic, renal, or psychiatric disorders
* Subject unable to follow the study during the 5 years of follow-up
* Subject in exclusion period of a previous study or simultaneously participating to any other clinical trial on metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-09; Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Type 2 Diabetes occurrence | 5 years (or less if occurrence of the condition)
  To understand the pathophysiological mechanisms involved in switching from pre-diabetes to type 2 diabetes and to identify new biomarkers of type 2 diabetes risk in this population

SECONDARY OUTCOMES:
Biomarkers | 7 to 10 years
  To highlight biomarkers of prediabetes, type 2 diabetes and cardiometabolic diseases, through genomics, proteomics and transcriptomics analyses performed on a biological sample collection.
Number of patients with pre-diabetes in North of France | 5 years
  To estimate the prevalence of prediabetes in the region Nord-Pas-de-Calais (France)
HbA1c measurement | 5 years
  To evaluate the role of HbA1c in screening for pre-diabetes and type 2 diabetes
Diabetes Risk Score | 5 years
  To assess the interest of Diabetes Risk Score (questionnaire used to evaluate a clinical risk) in identifying subjects at risk of type 2 diabetes
Others cardiovascular risk factors | 5 years
  To measure the prevalence of other cardiovascular risk factors observed along with prediabetes: dyslipidemia, metabolic hepatopathy

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Cariou, Pr., Principal Investigator — University Hospital of Nantes, France
Locations (1):
- Clinical Nutrition Center Naturalpha (CNCN), Lille, France

REFERENCES:
- [Derived] Croyal M, Wargny M, Chemello K, Chevalier C, Blanchard V, Bigot-Corbel E, Lambert G, Le May C, Hadjadj S, Cariou B. Plasma apolipoprotein concentrations and incident diabetes in subjects with prediabetes. Cardiovasc Diabetol. 2022 Feb 7;21(1):21. doi: 10.1186/s12933-022-01452-5. PMID 35130909
- [Derived] Wargny M, Smati S, Pichelin M, Bigot-Corbel E, Authier C, Dierry V, Zair Y, Jacquin V, Hadjadj S, Boursier J, Cariou B. Fatty liver index is a strong predictor of changes in glycemic status in people with prediabetes: The IT-DIAB study. PLoS One. 2019 Aug 29;14(8):e0221524. doi: 10.1371/journal.pone.0221524. eCollection 2019. PMID 31465427